CLINICAL TRIAL: NCT01262482
Title: A Phase 2 Trial of Oxaliplatin and Sorafenib Combination in Patients With Locally Advanced or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma, Relapsed After a Cisplatin Based Treatment
Brief Title: Study of Oxaliplatin and Sorafenib Combination to Treat Gastric Cancer Relapsed After a Cisplatin Based Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol Multidisciplinario del Cancer Digestivo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEMCAD-0802; 2008-004223-27 (EudraCT Number)
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2010-12

CONDITIONS: Advanced or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma (Relapsed After a Cisplatin Based Treatment)
Keywords: adenocarcinoma; gastric; gastroesophageal junction; Relapsed; sorafenib; oxaliplatin
MeSH Terms: conditions — Adenocarcinoma; Recurrence | interventions — Oxaliplatin; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxaliplatin + Sorafenib (Experimental)
  Interventions: Drug: Oxaliplatin; Drug: Sorafenib

INTERVENTIONS:
Drug: Oxaliplatin — 130 mg/m2, IV during 2 hours on day 1 of each 21 day cycle. Number of cycles: until progression, intolerance or unacceptable toxicity develops, or until patient or investigator decide to stop the treatment.
Drug: Sorafenib — 400mg, orally, 2 times per day. Until progression, intolerance or unacceptable toxicity develops, or until patient or investigator decide to stop the treatment.

SUMMARY:
In Spain, the gastric carcinoma is the 5th most frequent malignant tumor in women and the 6th in men, and represents the 3rd cause of cancer-related deaths amongst women and the 4th amongst men. The average of 5-year survival rate in Spain is under 30%. The main reason of it is that, despite carrying out an adjuvant treatment, more than the 50% will present relapsed disease.

Sorafenib has been the first RAF inhibitor, both of RAF-1 and B-rRAF and its b-RAF variant V600E. Moreover, it has shown its ability to inhibit other tyrosin-quinase receptors as VEGFR 2 and 3, c-kit, Flt-3 or PDGFR. Its activity has been clearly proven in clear cell renal carcinoma.

The mechanism by which Sorafenib seems to act is not because of the existence of a mutation of RAS or RAF, but because as there is a VHL shortage the HIP produces a VEGF, bFGF or TGF overexpression that produces in turn a hyper-stimulation on the RAF/ERK/MEK pathway.

The RAF/MEK/ERK pathway and angiogenesis seem to be clearly involved in the gastric carcinoma tumorigenesis and progression. Because of that, it seems interesting to associate Sorafenib to an oxaliplatin-based chemotherapy, which has shown its effectiveness in relapsed patients after receiving cisplatin-based schemes. Moreover, there is a phase 1 trial confirming the tolerance of the oxaliplatin and Sorafenib association, describing partial responses amongst gastric cancer patients previously treated with cisplatin.

ELIGIBILITY:
Inclusion Criteria:

1. Gastric or gastroesophageal junction adenocarcinoma confirmed by cytology or biopsy, with unresectable or metastatic disease which have progressed to a cisplatin-fluoropyrimidine based scheme (excluded neoadjuvant treatment administered with or without concomitant radiotherapy)
2. Older than 18 years at the moment of informed consent form signature
3. Age > 18 years
4. ECOG 0-2
5. Measurable disease by RECIST criteria. Lesions have to be measured by CT-scan or MRI
6. Life expectancy > 12 weeks
7. Adequate medullary reserve and hepatic and renal function, defined according to the following parameters:

   1. Hemoglobin ≥ 9g/dl
   2. Neutrophils ≥ 1,5 x 10^9/L
   3. Platelets ≥100 x 10^9/L
   4. Total bilirubin ≤ 1,5 times the upper limit of normal (ULN)
   5. ALT (GTP) and AST (GOT) ≤ 2,5 times the upper limit of normal (ULN) (≤ 5 times the ULN in patients with hepatic metastasis)
   6. PT-INR-PTT ≤ 1,5 times the ULN. (The patients under anticoagulant treatment with dicumarin or heparin can be included if there is no previous evidence of alteration in these parameters)
   7. Creatinine clearance > 30ml/min
8. The patients have to be able to understand the meaning of their participation in the trial and voluntary give their participation consent signing the informed consent form

Exclusion Criteria:

1. More than one line for the treatment of locally advanced disease
2. Active ischemic cardiopathy. History of cardiac disease defined as follow:

   1. Congestive cardiac failure > class 2 from the NYHA
   2. Active coronary disease. The recruitment of patients with solved myocardial infarction is allowed, if diagnosed at least 6 months before the trial start
   3. Cardiac arrhythmia requiring treatment with antiarrhythmic drugs. (The treatment with beta-adrenergic antagonists or digoxin is allowed)
   4. Non-controlled arterial hypertension
3. Non-controlled intercurrent illness
4. Symptomatic sensitive peripheral neuropathy
5. Another malignant disease diagnosed in the past 5 years, except in situ cervix carcinoma adequately treated, non-melanoma skin carcinoma, superficial bladder tumor (Ta, Tis and T1), or any tumor treated in a curative way until 3 years prior to the recruitment
6. Pregnant or breastfeeding women. Women will have to undergo a pregnancy test within 7 days prior to the recruitment. Both men and women recruited in the trial will have to use appropriate barrier contraceptive methods during their sexual relations during the trial period and at least until two weeks after its completion. Men participating in this trial will have to continue using this contraceptive methods at least until 3 months after the treatment completion
7. Chronic diseases: AIDS, Hepatitis B and/or Hepatitis C
8. Clinically active severe infection (Grade 2 NCI-CTC version 3.0)
9. Cerebral metastasis or meningeal tumor
10. Patients requiring chronic corticosteroid treatment or high doses of corticosteroids or any other immunosuppressive treatment
11. Patients having undergone a major surgery within the 4 weeks prior to the trial start
12. Patients having completed a chemotherapy or radiotherapy treatment within the 4 weeks prior to the clinical trial start (except palliative radiotherapy, within the 2-weeks prior to the clinical trial start)
13. Previous treatment using a RAS pathway inhibitor
14. Any medical or severe psychiatric condition or drug consumption involving a serious risk for the patient if taking part in the clinical trial or that can prevent the signature of the informed consent form
15. Patients unable to swallow medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-10; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival | anticipated 3 years
  Measurements according to RECIST criteria (Response Evaluation Criteria in Solid Tumors). Main techniques: CT-scan and Magnetic Resonance Imaging (MRI)

SECONDARY OUTCOMES:
Tumoral response | anticipated 3 years
  Measurements according to RECIST criteria (Response Evaluation Criteria in Solid Tumors). Main techniques: CT-scan and Magnetic Resonance Imaging (MRI)
Response duration | anticipated 3 years
  Duration of the partial or total response to the treatment. Evaluation and classification according to RECIST criteria (Response Evaluation Criteria in Solid Tumors)
Overall survival | anticipated 3 years
Toxicity | anticipated 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Marta Martin Richard, MD, Study Chair — Grupo Espanol Multidisciplinario del Cancer Digestivo
Locations (10):
- Spain (10):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Sant Pau, Barcelona
  - H. Josep Trueta, Girona
  - Centro Oncológico M.D. Anderson Spain, Madrid
  - Hospital de Fuenlabrada, Madrid
  - Hospital La Paz, Madrid
  - Hospital Althaia, Manresa
  - Clínica Universitaria de Navarra, Pamplona
  - Hospital Parc Taulí, Sabadell
  - Hospital General de Valencia, Valencia